CLINICAL TRIAL: NCT06405061
Title: A Prospective, Single-arm, Multicenter Phase II Clinical Study of Hepatic Arterial Perfusion Chemotherapy (FOLFOX) in Combination With Adebrelimab and Bevacizumab for Potentially Resectable Hepatocellular Carcinoma
Brief Title: Evaluation of Effectiveness and Safety of HAIC in Combination With Adebrelimab and Bevacizumab for Potentially Resectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-HCC-II-001
Record Dates: First submitted 2024-04-25; First posted 2024-05-08 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-04

CONDITIONS: Adebrelimab; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Adebrelimab: 1200 mg, IV, q3w Bevacizumab: 7.5 mg/kg, IV, q3w HAIC: (FOLFOX regimen:oxaliplatin 65 mg/m2, folinic acid 200 mg/m2, 5-Fu 200 mg/m2 push, followed by continuous infusion for 24h 1200 mg/m25-Fu), Q3W) every 3 weeks until 6 treatments have been completed or HAIC treatment is terminated when patients with fewer than 6 treatments develop intolerable adverse effects
  Interventions: Drug: Adebrelimab

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab: 1200 mg, IV, q3w
  Other Names: Bevacizumab; HAIC

SUMMARY:
Primary liver cancer mainly consists of three different pathologic types: hepatocellular carcinoma, intrahepatic cholangiocarcinoma, and hybrid HCC-ICC, of which HCC accounts for 90%. According to GLOBOCAN 2018 data, liver cancer is the sixth most prevalent tumor in the world, with about 841,100 new liver cancer cases and 781,600 deaths per year globally, which is the second leading cause of tumor deaths in men worldwide. China is a high incidence area of liver cancer, accounting for about 50% of the global incidence and deaths.

The treatment of HCC varies according to disease stage, which is based on the BCLC classification system, Child-Pugh liver function rating, and extent of disease. Approximately 30% of HCC cases are diagnosed in the early stages (i.e., BCLC stage 0 or A), and the main treatment options include surgical resection, ablation techniques, and liver transplantation. However, the 5-year recurrence rate remains as high as 70%. The recommended treatment for intermediate stage HCC (i.e., BCLC stage B) is hepatic artery intervention, i.e., transarterial chemoembolization (TACE), but the scope of applicability is limited due to concomitant disease and liver impairment factors, some patients do not derive a survival benefit from it, and patients ultimately progress after treatment and are no longer suitable for further TACE.

In recent years, the multi-drug combination therapy of systemic drugs combined with local therapy has also been gradually adopted, and studies have reported the feasibility of target drugs combined with ICI, TACE or HAIC for the treatment of unresectable hepatocellular carcinoma. The therapeutic aim of Adebrelimab (SHR-1316) is to inhibit tumor growth by specifically blocking the binding of PD-1 to PD-L1 and terminating the immunosuppressive signals generated by this receptor on T cells, so that T cells can re-recognize tumor cells and produce killing effects on them.

This study proposes an evaluation to explore the efficacy and safety of irinotecan liposome-based hepatic arterial perfusion chemotherapy (FOLFIRI) in combination with adebrelimab and bevacizumab for the treatment of potentially resectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. patients voluntarily enrolled in the study and signed an informed consent form.
2. 18-75 years old, both male and female.
3. patients with HCC diagnosed histologically, cytologically, or clinically.
4. CNLC-IIb to IIIaHCC (IIIa is limited to combined portal vein branch thrombosis Ching's staging grade I/II) of the Guidelines for the Management of Primary Liver Cancer (2022 edition).
5. not have received any prior local and systemic therapy for HCC.
6. at least one measurable lesion (the measurable lesion is ≥10 mm in long diameter or ≥15 mm in short diameter of enlarged lymph node on spiral CT scan according to RECISTv1.1).
7. Child-Pugh score ≤7.
8. ECOG score:0~1.
9. Expected survival ≥12 weeks.
10. Vital organs function in accordance with the following requirements (within 7 days prior to initiation of study treatment).

(1) Routine blood tests: (except hemoglobin, which has not been transfused, granulocyte colony-stimulating factor [G-CSF], or corrected with medication within 14 days prior to screening): absolute neutrophil count ≥ 1.5 x 109/L; platelets ≥ 75 x 109/L; hemoglobin ≥ 90 g/L.

(2) Biochemical tests: (no albumin transfusion within 14 days prior to screening): serum albumin ≥29g/L; serum total bilirubin ≤1.5×upper limit of normal range (ULN); alanine aminotransferase (ALT), aspartate aminotransferase acid enzyme (AKP) ≤5×ULN; serum creatinine (Cr) ≤1.5ULN or Cr clearance >50mL/min.

(3) International normalized ratio (INR) ≤ 2.3 or prothrombin time (PT) exceeding the range of normal control ≤ 6 seconds.

(4) Urine protein <2+ (if urine protein ≥2+, 24-hour (h) urine protein quantification can be performed, and 24-h urine protein quantification <1.0 g can be enrolled).

11. If the patient has active hepatitis B virus (HBV) infection: HBV-deoxyribonucleic acid (DNA) must be <500 IU/mL (or <2500 copies/mL if only copies/mL are available at the study center), and has received at least 14 days of anti-HBV treatment prior to the initiation of study treatment (based on the standard of care in the local area, e.g., entecavir) and is willing to be enrolled at the time of study treatment. Patients who are hepatitis C virus (HCV) ribonucleic acid (RNA)-positive must be receiving antiviral therapy according to standard local treatment guidelines and have liver function within CTCAE grade 1 elevation.

12. Patients must agree to use contraception for at least 120 days from the date of informed consent until the last dose of study drug. Must have had a negative serum HCG test within 7 days prior to starting study treatment; must not be breastfeeding.

Exclusion Criteria:

1. Known hepatobiliary ductal cell carcinoma, sarcomatoid HCC, mixed cell carcinoma and fibrous platysmal cell carcinoma; active malignant tumors other than HCC within 5 years or at the same time. Cured limited tumors, such as basal cell carcinoma of the skin, squamous carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, carcinoma in situ of the breast, etc. can be enrolled.
2. Patients with combined portal vein branch thrombosis of grade III or above in Cheng's staging.
3. Patients who are going to undergo or have previously undergone organ or allogeneic bone marrow transplantation.
4. Patients with clinically symptomatic moderate or severe ascites that requires therapeutic puncture or drainage or Child-Pugh score >2 (except those with only a small amount of ascites on imaging but not accompanied by clinical symptoms); uncontrolled or moderate amount or more of pleural effusion or pericardial effusion.
5. Esophageal varices or fundal bleeding due to portal hypertension within the past 6 months; Presence of severe (G3) varices detected by endoscopy 3 months prior to initial dosing; Evidence of portal hypertension (including imaging findings of spleen more than 10 cm in length and platelets less than 100) and high risk of bleeding as assessed by the investigator.
6. Arteriovenous thromboembolic events within the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other history of severe thromboembolism. Implantable IV port or catheter derived thrombosis, or superficial vein thrombosis, except for thrombus stabilization after routine anticoagulation therapy.
7. Known hereditary or acquired bleeding (e.g., coagulation disorders) or thrombotic tendencies, such as in patients with hemophilia; Currently using or have recently (within 10 days prior to initiation of study treatment) used for therapeutic purposes full-dose oral or injectable anticoagulant or thrombolytic medications (prophylactic use of low-dose aspirin, low molecule heparin is permitted).
8. current or recent (within 10 days prior to start of study treatment) treatment with aspirin (>325 mg/day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel and cilostazol.
9. Thrombotic or embolic events, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc., within 6 months prior to the start of study treatment.
10. Uncontrolled cardiac clinical symptoms or diseases, such as: (1) Class II or higher cardiac insufficiency according to the New York Heart Association (NYHA) criteria (see Annex 5) or cardiac ultrasound: LVEF (left ventricular ejection fraction) < 50%; (2) unstable angina pectoris; (3) myocardial infarction within 1 year prior to the start of the study; (4) clinically significant supraventricular or ventricular arrhythmia requiring a cardiovascular or cardioembolic intervention; and (5) clinically significant supraventricular or ventricular arrhythmia requiring a cardiovascular or cardiac intervention; (6) cardiac disease or disease of the heart. or ventricular arrhythmia requiring treatment or intervention; (5) QTc>450ms (men); QTc>470ms (women) (QTc intervals were calculated using the Fridericia formula; if the QTc was abnormal, three consecutive tests were performed at 2-minute intervals, and the average value was taken).
11. have hypertension that is not well controlled by antihypertensive medication (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg) (based on the average of ≥2 BP readings), allowing the achievement of the above parameters through the use of antihypertensive therapy; have had a previous hypertensive crisis or hypertensive encephalopathy.
12. significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to the start of study treatment; and
13. severe, unhealed or gaping wounds and active ulcers or untreated fractures.
14. major surgical treatment (other than diagnostic) within 4 weeks prior to the start of study treatment or anticipated need for major surgical treatment during the study period.
15. previous intestinal obstruction and/or previous clinical signs or symptoms of gastrointestinal obstruction within 6 months prior to initiation of study treatment, including incomplete obstruction related to a pre-existing condition or requiring routine parenteral hydration, parenteral nutrition, or tube feeding/tube feeding.
16. Patients may be enrolled in the study if at the time of initial diagnosis patients with incomplete obstruction/obstruction syndrome/signs/symptoms of intestinal obstruction receive definitive (surgical) treatment to abate symptoms.
17. evidence of an intra-abdominal pneumoperitoneum that cannot be explained by puncture or recent surgery.
18. previous or current central nervous system metastases.
19. Metastatic disease involving major airways or blood vessels (e.g., complete occlusion of the portal trunk or vena cava due to tumor invasion, which refers to the confluence of the splenic vein and the superior mesenteric vein, and the division of the hepatic portal vein into right and left branches) or a centrally located large mediastinal tumor mass (<30 mm from the crista longitudinalis).
20. those with a history of hepatic encephalopathy.
21. current concomitant interstitial pneumonia or interstitial lung disease, or a previous history of interstitial pneumonia or interstitial lung disease requiring hormonal therapy, or other conditions that may interfere with the determination and management of immune-related pulmonary toxicity such as pulmonary fibrosis, organic pneumonia (e.g., occlusive bronchiectasis), pneumoconiosis, drug-associated pneumonia, idiopathic pneumonia, or active pneumonia as seen on a screening chest computed tomography (CT) picture Evidence or severely impaired lung function in subjects with a history of radiation pneumonitis in the permitted radiation field; active tuberculosis.
22. presence of active autoimmune disease or history of autoimmune disease with potential for relapse (including, but not limited to: autoimmune hepatitis, interstitial pneumonitis, uveitis, enterocolitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects who can be controlled by hormone replacement therapy only are eligible for enrollment]); subjects with skin conditions that do not require systemic treatment such as vitiligopsoriasis, alopecia areata, controlled type I diabetes mellitus treated with insulin or asthma that has completely resolved in childhood and does not require any intervention in adulthood may be included; asthmatics requiring medical intervention with bronchodilators may not be included.
23. Immunosuppressive or systemic hormone therapy for immunosuppression within 14 days prior to initiation of study treatment (dose >10 mg/day prednisone or other equipotent hormone).
24. Use of strong CYP3A4/CYP2C19 inducers including rifampicin (and its analogs) and oncolytic or strong CYP3A4/CYP2C19 inhibitors within 14 days prior to initiation of study treatment.
25. severe infection within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia; therapeutic antibiotics given orally or intravenously within 2 weeks prior to initiation of study treatment (patients receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection or exacerbation of COPD are eligible for study participation).
26. Patients with congenital or acquired immune deficiency (e.g., HIV-infected patients).
27. Combined hepatitis B and hepatitis C co-infection.
28. Use of immunosuppressive drugs within 4 weeks prior to the first dose; and
29. Received live attenuated vaccine within 4 weeks prior to the first dose or plan to receive live attenuated vaccine during the study.
30. Received a traditional Chinese medicine with an antitumor indication or a drug with immunomodulatory effects within 2 weeks prior to the first dose of study drug.
31. previous treatment with other anti-PD-1 antibodies or other immunotherapy targeting PD-1/PD-L1.
32. palliative radiotherapy to non-target lesions for symptom control is permitted and must have been completed at least 2 weeks prior to the initiation of study treatment use, with no recovery from radiotherapy-induced adverse events to ≤ CTCAE grade 1.
33. have received other experimental drug therapy within 28 days prior to initiation of study treatment.
34. In the judgment of the investigator, the patient has other factors that may affect the results of the study or cause this study to be forced to be terminated in midstream, such as alcoholism, drug abuse, other serious illnesses (including psychiatric illnesses) that require comorbid treatment, serious laboratory test abnormalities, accompanied by family or social factors that would affect the patient's safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate per RECIST 1.1 | From treatment initiation to progressive disease or EOT due to any cause, assessed up to 1 year
  Defined as proportion of patients who have a best response of CR or PR

SECONDARY OUTCOMES:
Major Pathological response | After surgical excision with follow up of an average of 1 year
  the percentage of tumor cells before and after treatment was compared according to biopsy specimens before neoadjuvant therapy and pathological specimens after surgery; the percentage of tumor cells was evaluated on resected tumor slides. MPR was defined as ≤ 10% tumor cells.
Disease Control Rate | From treatment initiation to progressive disease or EOT due to any cause, assessed up to 1 year
  Defined as proportion of patients who have CR or PR or SD
R0 resection rate | After surgical excision with follow up of an average of 1 year
  Patients who underwent radical resection as a percentage of the total number of patients who underwent surgical resection
Pathological complete response | After surgical excision with follow up of an average of 1 year
  Disappearance of tumor cells from resected specimen
Event Free Survival | From treatment initiation to progressive disease, discontinuation of the treatment for any reason, or death due to any cause, assessed up to 1 year
  From date of surgery until the date of recurrence detection.
Overall survival | From treatment initiation until death due to any cause, assessed up to 3 year
  Defined as the time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Third Central Hospital of Tianjin, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
Study protocol